CLINICAL TRIAL: NCT04628078
Title: LAAC-registry: Clinical Outcome After Echocardiography-guided LAA-closure
Status: Recruiting | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Other Study IDs: 2016-01742
Record Dates: First submitted 2020-11-05; First posted 2020-11-13 (Actual); Last update posted 2023-02-22 (Actual); Status verified 2023-02

CONDITIONS: Atrial Fibrillation; Cardiovascular Diseases; Thromboembolism
Keywords: Left atrial appendage closure; Amulet; Watchman; Watchman flx; Acp; Cardiac computed tomography angiography; Transesophageal echocardiography; Peridevice leak; Thromboembolic events; Atrial fibrillation
MeSH Terms: conditions — Atrial Fibrillation; Cardiovascular Diseases; Thromboembolism; Cerebral Palsy, Ataxic, Autosomal Recessive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Use of echocardiography guidance for LAAC — Since August 2015, the echocardiography is routinely used by majority of operators to guide LAAC

SUMMARY:
The study aims at comparing, in a large cohort of consecutive clinically indicated left atrial appendage closure, clinical and imaging outcomes between different subpopulations.

DETAILED DESCRIPTION:
Percutaneous left atrial appendage closure (LAAC) has established itself in clinical practice as a safe and efficient therapeutic option for atrial fibrillation patients with a relative/absolute contraindication to oral anticoagulation. The purpose of this observational study is to prospectively collect procedural and follow-up data of all patients submitted to a clinically indicate LAAC in order to assess the impact of patient characteristics, procedural technique (imaging used to guide/plan procedure, device implanted, post-procedural drug regimens, etc.) on procedural safety and efficacy. The endpoints will be assessed by means of clinical follow-up at 1-3-5 years after LAAC and imaging exams (TEE at1-3 months, CCTA at 1-13months).

ELIGIBILITY:
Inclusion Criteria:

* Age> 18
* Written informed consent to participate in the study
* Patients with paroxysmal, persistent, or permanent non-valvular AF and CHA2DS2-VASc Score of ≥2 that are planned for an elective LAA-closure
* Anatomic characteristics allow placement of a CE marked device, dedicated for LAAC

Exclusion Criteria:

* None. Considering the nature of the project, which is to prospectively collect information on all patients treated with LAAC in our center, we will only exclude patients unwilling to sign the informed consent.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with paroxysmal, persistent, or permanent non-valvular AF and CHA2DS2-VASc Score of ≥2 that are scheduled to undergo to an elective Left Atrial Appendage Closure
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2015-08-12 (Actual); Primary Completion 2023-06-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Primary Safety Endpoint | 7 days
  Composite of Death, cerebrovascular events, cardiac tamponade, need for urgent surgery, need for cardiopulmonary resuscitation, device embolization, non vascular access-related major or life-threatening bleeding (according to the Bleeding academic research Criteria (BARC) type 3a, 3b, 3c, or 5) or acute kidney injury.
Primary Efficacy Endpoint - Incidence of cardiovascular death, ischemic stroke and systemic embolism | 1 to 5 Years
  Protection from cardiovascular death, ischemic stroke and systemic embolism
Secondary Efficacy Endpoint - Incidence of technical success | 7 days to 13 months
  Technical success defined as adequate LAA ostium closure (without residual PDL>5mm or patent lobes) in absence of device complications (according to the Munich Consensus Document)
Feasibility Endpoint - Total procedure time (min) | During the LAAC Procedure (≃ 60 minutes )
  Total procedure time (min)
Feasibility Endpoint - dose of contrast medium (ml) | During the LAAC Procedure (≃ 60 minutes )
  dose of contrast medium (ml)
Feasibility Endpoint - dose of x-ray (cGy.cm2) | During the LAAC Procedure (≃ 60 minutes )
  dose of x-ray (cGy.cm2)
Feasibility Endpoint - number of device implantation attempt during the procedure (number) | During the LAAC Procedure (≃ 60 minutes )
  number of device implantation attempt during the procedure (number)
Feasibility Endpoint - number of device change during the procedure (number) | During the LAAC Procedure (≃ 60 minutes )
  number of device change during the procedure (number)
Net Clinical Benefit Endpoint | 1 to 5 years
  Composite of death, stroke, systemic embolism, pulmonary embolism, myocardial infarction, and major or life-threatening bleeding (according to the Bleeding academic research Criteria (BARC) type 3a, 3b, 3c, or 5) not procedure-related.
LAA patency | 45 days to 13 months
  LAA patency and its subtypes as evaluated by TEE and/or CCTA
Device related thrombus | 45 days to 13months
  Device related thrombus detected by TEE and /or CCTA on the atrial surface of device

SECONDARY OUTCOMES:
Percentage of atrial surface of device covered | 45 days - 3 months - 13months
  % (device sealing surrogate)
Maximal Hypoattentuated Thickening on atrial surface of device | 45 days - 3 months - 13months
  mm (device sealing surrogate)
Percentage of device length coverage | 45 days - 3 months - 13months
  % (device sealing surrogate)

CONTACTS AND LOCATIONS:
Overall Officials: Lorenz Räber, Prof., Principal Investigator — Insel Gruppe AG, Inselspital, Universitätsklinik für Kardiologie
Locations (1):
- Bern University Hospital Inselspital, Bern, Switzerland

REFERENCES:
- [Background] Go AS, Mozaffarian D, Roger VL, Benjamin EJ, Berry JD, Blaha MJ, Dai S, Ford ES, Fox CS, Franco S, Fullerton HJ, Gillespie C, Hailpern SM, Heit JA, Howard VJ, Huffman MD, Judd SE, Kissela BM, Kittner SJ, Lackland DT, Lichtman JH, Lisabeth LD, Mackey RH, Magid DJ, Marcus GM, Marelli A, Matchar DB, McGuire DK, Mohler ER 3rd, Moy CS, Mussolino ME, Neumar RW, Nichol G, Pandey DK, Paynter NP, Reeves MJ, Sorlie PD, Stein J, Towfighi A, Turan TN, Virani SS, Wong ND, Woo D, Turner MB; American Heart Association Statistics Committee and Stroke Statistics Subcommittee. Heart disease and stroke statistics--2014 update: a report from the American Heart Association. Circulation. 2014 Jan 21;129(3):e28-e292. doi: 10.1161/01.cir.0000441139.02102.80. Epub 2013 Dec 18. No abstract available. PMID 24352519
- [Background] Feigin VL, Forouzanfar MH, Krishnamurthi R, Mensah GA, Connor M, Bennett DA, Moran AE, Sacco RL, Anderson L, Truelsen T, O'Donnell M, Venketasubramanian N, Barker-Collo S, Lawes CM, Wang W, Shinohara Y, Witt E, Ezzati M, Naghavi M, Murray C; Global Burden of Diseases, Injuries, and Risk Factors Study 2010 (GBD 2010) and the GBD Stroke Experts Group. Global and regional burden of stroke during 1990-2010: findings from the Global Burden of Disease Study 2010. Lancet. 2014 Jan 18;383(9913):245-54. doi: 10.1016/s0140-6736(13)61953-4. PMID 24449944
- [Background] Gloekler S, Meier B, Windecker S. Left atrial appendage closure for prevention of cardioembolic events. Swiss Med Wkly. 2016 May 31;146:w14298. doi: 10.4414/smw.2016.14298. eCollection 2016. PMID 27244534
- [Background] Blackshear JL, Odell JA. Appendage obliteration to reduce stroke in cardiac surgical patients with atrial fibrillation. Ann Thorac Surg. 1996 Feb;61(2):755-9. doi: 10.1016/0003-4975(95)00887-X. PMID 8572814
- [Background] Holmes DR Jr, Doshi SK, Kar S, Price MJ, Sanchez JM, Sievert H, Valderrabano M, Reddy VY. Left Atrial Appendage Closure as an Alternative to Warfarin for Stroke Prevention in Atrial Fibrillation: A Patient-Level Meta-Analysis. J Am Coll Cardiol. 2015 Jun 23;65(24):2614-2623. doi: 10.1016/j.jacc.2015.04.025. PMID 26088300
- [Background] Reddy VY, Sievert H, Halperin J, Doshi SK, Buchbinder M, Neuzil P, Huber K, Whisenant B, Kar S, Swarup V, Gordon N, Holmes D; PROTECT AF Steering Committee and Investigators. Percutaneous left atrial appendage closure vs warfarin for atrial fibrillation: a randomized clinical trial. JAMA. 2014 Nov 19;312(19):1988-98. doi: 10.1001/jama.2014.15192. PMID 25399274
- [Background] Holmes DR Jr, Kar S, Price MJ, Whisenant B, Sievert H, Doshi SK, Huber K, Reddy VY. Prospective randomized evaluation of the Watchman Left Atrial Appendage Closure device in patients with atrial fibrillation versus long-term warfarin therapy: the PREVAIL trial. J Am Coll Cardiol. 2014 Jul 8;64(1):1-12. doi: 10.1016/j.jacc.2014.04.029. PMID 24998121
- [Background] Koskinas KC, Shakir S, Fankhauser M, Nietlispach F, Attinger-Toller A, Moschovitis A, Wenaweser P, Pilgrim T, Stortecky S, Praz F, Raber L, Windecker S, Meier B, Gloekler S. Predictors of Early (1-Week) Outcomes Following Left Atrial Appendage Closure With Amplatzer Devices. JACC Cardiovasc Interv. 2016 Jul 11;9(13):1374-83. doi: 10.1016/j.jcin.2016.04.019. PMID 27388826
- [Background] Holmes DR, Reddy VY, Turi ZG, Doshi SK, Sievert H, Buchbinder M, Mullin CM, Sick P; PROTECT AF Investigators. Percutaneous closure of the left atrial appendage versus warfarin therapy for prevention of stroke in patients with atrial fibrillation: a randomised non-inferiority trial. Lancet. 2009 Aug 15;374(9689):534-42. doi: 10.1016/S0140-6736(09)61343-X. PMID 19683639
- [Background] Kappetein AP, Head SJ, Genereux P, Piazza N, van Mieghem NM, Blackstone EH, Brott TG, Cohen DJ, Cutlip DE, van Es GA, Hahn RT, Kirtane AJ, Krucoff MW, Kodali S, Mack MJ, Mehran R, Rodes-Cabau J, Vranckx P, Webb JG, Windecker S, Serruys PW, Leon MB. Updated standardized endpoint definitions for transcatheter aortic valve implantation: the Valve Academic Research Consortium-2 consensus document. Eur Heart J. 2012 Oct;33(19):2403-18. doi: 10.1093/eurheartj/ehs255. PMID 23026477
- [Background] Mehran R, Rao SV, Bhatt DL, Gibson CM, Caixeta A, Eikelboom J, Kaul S, Wiviott SD, Menon V, Nikolsky E, Serebruany V, Valgimigli M, Vranckx P, Taggart D, Sabik JF, Cutlip DE, Krucoff MW, Ohman EM, Steg PG, White H. Standardized bleeding definitions for cardiovascular clinical trials: a consensus report from the Bleeding Academic Research Consortium. Circulation. 2011 Jun 14;123(23):2736-47. doi: 10.1161/CIRCULATIONAHA.110.009449. No abstract available. PMID 21670242
- [Background] Tzikas A, Holmes DR Jr, Gafoor S, Ruiz CE, Blomstrom-Lundqvist C, Diener HC, Cappato R, Kar S, Lee RJ, Byrne RA, Ibrahim R, Lakkireddy D, Soliman OI, Nabauer M, Schneider S, Brachmann J, Saver JL, Tiemann K, Sievert H, Camm AJ, Lewalter T. Percutaneous left atrial appendage occlusion: the Munich consensus document on definitions, endpoints, and data collection requirements for clinical studies. Europace. 2017 Jan;19(1):4-15. doi: 10.1093/europace/euw141. Epub 2016 Aug 18. PMID 27540038
- [Derived] Galea R, Bini T, Krsnik JP, Touray M, Temperli FG, Kassar M, Papadis A, Gloeckler S, Brugger N, Madhkour R, Seiffge DJ, Roten L, Siontis GCM, Heg D, Windecker S, Raber L. Pericardial Effusion After Left Atrial Appendage Closure: Timing, Predictors, and Clinical Impact. JACC Cardiovasc Interv. 2024 Jun 10;17(11):1295-1307. doi: 10.1016/j.jcin.2024.01.310. Epub 2024 May 22. PMID 38795087